CLINICAL TRIAL: NCT06693401
Title: Forensic Analysis of Dynamic Handwriting Characteristics After Rehabilitation Intervention in People with Parkinson's Disease - Pilot Study
Brief Title: Forensic Handwriting Analysis in People with Parkinson's Disease - Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Egas Moniz - Cooperativa de Ensino Superior, CRL (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1171/23ParkinsonHandwriting
Record Dates: First submitted 2024-05-02; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Parkinson Disease
Keywords: Forensic Characterization; Occupational Therapy; Physiotherapy; Graphoscopic Assessment; Dynamic Features
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Physiotherapy Intervention rehabilitation program was implemented in both study groups in accordance to the usual physiotherapeutic rehabilitation approach through a programme according to the European and American Guidelines for Physical Therapy in Parkinson's Disease, with the purpose of improving balance and reducing the risk of falls, enhancing mobility and motor function, managing muscle stiffness and rigidity, addressing gait abnormalities, and providing education and support.
  Occupational Therapy rehabilitation program was implemented only in the Intervention Group, through handbooks for handwriting occupational therapy exercises in Portuguese language, with exercises to be performed for about 45 minutes, three times a week. Each participant was offered a kit with all the materials needed to perform the handwriting and fine motor skills exercises (1 ping-pong ball, 1 anti-stress ball, 1 plastic coin, 2 rubber bands, 2 beans and 10 paper clips).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Physiotherapy programme (Active Comparator): The active comparator arm consisted of implementing the conventional physiotherapy programme in accordance to the usual physiotherapeutic rehabilitation approach through a programme tailored to the specific difficulties of each individual and adapted to their needs on a session-by-session basis and framed according the European and American Guidelines for Physical Therapy in Parkinson's Disease.
  Interventions: Other: Control Group: conventional physiotherapy programme
- Physiotherapy programme + Occupational Therapy programme (Experimental): The experimental arm consisted of adding an occupational therapy programme to the conventional physiotherapy programme. The occupational therapy intervention consisted in fine motor tasks exercises implemented to address hand dexterity by training hand function with a range of exercises that enhance the main skills that make our hands useful and functional, such as object manipulation, finger isolation, finger and hand extension and flexion, and coordination and handwriting exercises in Portuguese language.
  Interventions: Other: Intervention group: PD rehabilitation complemented with Occupational Therapy programme

INTERVENTIONS:
Other: Intervention group: PD rehabilitation complemented with Occupational Therapy programme — In intervention group both Physiotherapy and Occupational Therapy programmes were implemented.
  Occupational Therapy programme consisted in trainning the amplitude of the movements involved in the realization of each letter of the alphabet separately and through fine motor exercises. Specifically the tasks consisted of performing:
  1. 2 types of handwriting exercises, namely for tracing the upper and lower-case letters of the alphabet guided by dotted lines and writing a sentence with and without spatial boundaries, in Portuguese language (to be performed for about 45 minutes, three times a week) and;
  2. 4 groups of fine motor tasks exercises, namely for hand manipulation (2 exercises), finger isolation (3 exercises), finger flexion and extension (2 exercises) and coordination (1 exercise). All exercises were performed 10 times, in triplicate, for each hand on a regular basis of 2-3 times per week.
  Arms: Physiotherapy programme + Occupational Therapy programme
Other: Control Group: conventional physiotherapy programme — In this group only the conventional physiotherapy programme was implemented. This programme has the purpose of improving balance and reducing the risk of falls, enhancing mobility and motor function, managing muscle stiffness and rigidity, addressing gait abnormalities, and providing education and support. In this regard, participants were guided and supervised in each physiotherapy session by a Parkinson's disease healthcare specialist.
  Arms: Physiotherapy programme

SUMMARY:
Graphoscopic analysis of handwriting is influenced by various internal and external factors, and individuals with degenerative diseases like Parkinson's face challenges due to limitations in motor abilities, impacting Instrumental Activities of Daily Living (IADL) such as handwriting skills. The absence of encouraging outcomes from interventions in handwriting rehabilitation programs and graphoscopic assessment tools, persists as an ongoing challenge.

This pilot study undertook an investigation into the forensic characterization of handwriting in people with Parkinson's Disease (PD). The main goal was to evaluate and compare the effect of 2 rehabilitation programs on handwriting, particularly, regarding 9 static and dynamic features, in individuals with PD.

Additionally, this study contributed to the development of a comprehensive protocol, incorporating the most suitable and discriminatory clinical and graphoscopic assessment tools in the context of PD, and to formulate an occupational therapy rehabilitation program focused on enhancing the dexterity and fine motor skills of the upper limbs, crucial for improved performance in Instrumental Activities of Daily Living (IADLs).

The pilot trial involved two groups: an intervention group (IG) undergoing traditional physiotherapy and occupational therapy programs (TPRP + OTRP), and a control group (CG) undergoing traditional physiotherapy alone (TPRP).

The objective was to characterize and compare handwriting before and after the rehabilitation programs.

Participants underwent assessments at the study's commencement and after 12 weeks of intervention. Graphoscopic assessment utilized a Wacom One DTC133W0A tablet and NeuroScript's v6.1 MovAlyzeR software. Clinical assessments included the Jebsen Taylor Hand Function Test, Movement Disorder Society Unified Parkinson Disease Rate Scale, and the Parkinson Disease Questionnaire 8 tests.

DETAILED DESCRIPTION:
The potential participants were recruited through the Clínica Neurovida and Clínica de Fisioterapia Egas Moniz (Monte da Caparica) who, on their own initiative, start attending the partner institutions or are members. People who meet the eligibility criteria, after initial clinical diagnosis, were invited to participate in this study. Before entering the clinical trial, participants were fully briefed on the conditions under which they underwent during the tests and rehabilitation program procedures, after which a consent informed form was signed for the use of these results for research purposes. The collection, processing and dissemination of data were carried out anonymously.

Both intervention programs were performed during 12 weeks.

* Traditional physiotherapy rehabilitation program (TPRP) (practice for 1h, twice a week) - implemented according to the European Physiotherapy Guideline for Parkinson's Disease.
* Occupational therapy rehabilitation program (OTRP) - implemented through workbooks, practice for 30 min, three times a week, according to the Guidelines for Occupational Therapy in Parkinson's Disease Rehabilitation.

The motor tasks for the OTRP consists in performing, 2-3 times a week, exercises included in a workbook (drawing the upper and lower case letters of the alphabet guided by dotted lines, writing a sentence with and without spatial limits) and performing 3 groups of fine motor tasks: Hand manipulation (2 exercises), Finger isolation (3 exercises), Finger flexion and extension (2 exercises) and Coordination (1 exercise). All exercises should be performed 10 times, in triplicate, for each hand. Subjects evaluate the subjective performance of the execution through a questionnaire at the end of each exercise where they indicate whether they performed fully, partially or not at all.

Handwriting Sample collection In the first stage, the participants of this pilot trial were asked to perform specific motor tasks (estimated time -15 min) by the researcher responsible for sample collection, directly on the surface of a digitizer (Wacom One 13'), using an appropriate stylus and capturing software (MovAlyzeR v6.1 - NeuroScript) (t0). These samples were adequately identified and conditioned. After assessment (t0), both groups (control and intervention) were submitted to a rehabilitation intervention, followed by handwriting assessments after 12 weeks (t1) of rehabilitation interventions. Dynamic features (e.g.: average pen pressure, normalized jerk, duration, horizontal size, vertical size, relative pen down duration, number of acceleration peaks, average absolute velocity and absolute size) were extracted and compared from the digital samples collected before (t0) and after the rehabilitation intervention (t1).

Motor function assessment Assessment of motor function were performed in the 2 evaluation moments (t0, t1): upper limb throughout MDS UPDRS (2.7, 3.3.b, 3.3c, 3.4.a, 3.4.b, 3.5.a, 3.5.b, 3.6.a, 3.6.b) and Jebsen-Taylor tests.

ELIGIBILITY:
Inclusion Criteria:

* individuals with an early to middle diagnosis of PD stage 2-3 on the Hoehn and Yahr scale
* level of education from the fourth grade onwards
* Portuguese as their native language.

Exclusion Criteria:

* presence of physical or mental pathologies or clinical conditions other than PD that may impact writing or the nervous system
* color blindness
* deafness
* thyroid gland dysfunctions.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-03-14 (Actual); Primary Completion 2023-07-21 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Absolute Size | Implemented at baseline (T0) and after 12 weeks of intervention (T1)
  Absolute Size (pt - point, 1/72 of an inch) was assessed through Graphoscopic assessment for each exercise: drawing a narrow Archimedean spiral (SSD), drawing a wide Archimedean spiral (SLD) , drawing two overlapping regular pentagons (PTG), and writing a sentence (WRI) "Os peixes retiram o ar da água" (Fish extract air out of water).
Horizontal Size (HS) | Implemented at baseline (T0) and after 12 weeks of intervention (T1)
  Horizontal Size (pt - point, 1/72 of an inch) was assessed through Graphoscopic assessment for each exercise: drawing a narrow Archimedean spiral (SSD), drawing a wide Archimedean spiral (SLD) , drawing two overlapping regular pentagons (PTG), and writing a sentence (WRI) "Os peixes retiram o ar da água" (Fish extract air out of water).Implemented at baseline (T0) and after 12 weeks of intervention (T1)
Vertical Size | Implemented at baseline (T0) and after 12 weeks of intervention (T1)
  Vertical Size (pt - point, 1/72 of an inch) was assessed through Graphoscopic assessment for each exercise: drawing a narrow Archimedean spiral (SSD), drawing a wide Archimedean spiral (SLD) , drawing two overlapping regular pentagons (PTG), and writing a sentence (WRI) "Os peixes retiram o ar da água" (Fish extract air out of water).
Average Absolute Velocity | Implemented at baseline (T0) and after 12 weeks of intervention (T1)
  Average Absolute Velocity (pt/s ) was assessed through Graphoscopic assessment for each exercise: drawing a narrow Archimedean spiral (SSD), drawing a wide Archimedean spiral (SLD) , drawing two overlapping regular pentagons (PTG), and writing a sentence (WRI) "Os peixes retiram o ar da água" (Fish extract air out of water).
Duration | Implemented at baseline (T0) and after 12 weeks of intervention (T1)
  Duration (s) was assessed through Graphoscopic assessment for each exercise: drawing a narrow Archimedean spiral (SSD), drawing a wide Archimedean spiral (SLD) , drawing two overlapping regular pentagons (PTG), and writing a sentence (WRI) "Os peixes retiram o ar da água" (Fish extract air out of water).
Relative Pen-Down Duration | Implemented at baseline (T0) and after 12 weeks of intervention (T1)
  Relative Pen-Down Duration (s) was assessed through Graphoscopic assessment for each exercise: drawing a narrow Archimedean spiral (SSD), drawing a wide Archimedean spiral (SLD) , drawing two overlapping regular pentagons (PTG), and writing a sentence (WRI) "Os peixes retiram o ar da água" (Fish extract air out of water).
Average Pen Pressure | Implemented at baseline (T0) and after 12 weeks of intervention (T1)
  Average Pen Pressure (g) was assessed through Graphoscopic assessment for each exercise: drawing a narrow Archimedean spiral (SSD), drawing a wide Archimedean spiral (SLD) , drawing two overlapping regular pentagons (PTG), and writing a sentence (WRI) "Os peixes retiram o ar da água" (Fish extract air out of water).
Normalized Jerk | Implemented at baseline (T0) and after 12 weeks of intervention (T1)
  Normalized Jerk (m/s^3) was assessed through Graphoscopic assessment for each exercise: drawing a narrow Archimedean spiral (SSD), drawing a wide Archimedean spiral (SLD) , drawing two overlapping regular pentagons (PTG), and writing a sentence (WRI) "Os peixes retiram o ar da água" (Fish extract air out of water).
Parkinson Disease Questionnaire 8 (PDQ-8) | Implemented at baseline (T0) and after 12 weeks of intervention (T1)
  Parkinson Disease Questionnaire 8 (score: range from 0 to 32 points) was assessed through clinical assessment and is a simplified tool derived from the PDQ-39 questionnaire, which assesses the overall well-being of an individual with Parkinson's disease (PD).
Movement Disorder Society Unified Parkinson Disease Rating Scale (MDS-UPDRS) | Implemented at baseline (T0) and after 12 weeks of intervention (T1)
  Movement Disorder Society Unified Parkinson Disease Rating Scale (MDS-UPDRS) (score: range from 0 to 26 points) was assessed through clinical assessment and is a comprehensive scale that evaluates both motor and non-motor symptoms of PD. In this particular study, the following subgroupsof the Official MDS UPDRS Portuguese Translation were considered: Writing (item 2.7); Bradykinesia (items 3.4, 3.5 and 3.6) and Tremor (items 3.15, 3.16 and 3.17).
Jebsen-Taylor Hand Function Test (JTHFT) | Implemented at baseline (T0) and after 12 weeks of intervention (T1)
  Jebsen-Taylor Hand Function Test (JTHFT) (s) was assessed through clinical assessment and is a tool commonly used by occupational therapists to characterize manual function in individuals with PD. This test evaluates the time taken to complete 7 exercises with the left and right hand. The mean reference subtest scores are considered for women and men, stratified by age groups (20-59 years and 60-94), and presented for both dominant and non-dominant hands.

SECONDARY OUTCOMES:
Age | At baseline
  Sample characterisation (years)
Gender | At baseline
  Sample percentual gender characterisation (male/female/other)
Years of Parkinson Disease | At baseline
  Sample characterisation (years)

CONTACTS AND LOCATIONS:
Locations (1):
- Egas Moniz School of Health and Science, Almada, Monte de Caparica, Portugal